CLINICAL TRIAL: NCT06163924
Title: To Investigate the Effect of Multidisciplinary Care Approach on Cardiovascular Risk Modification in Prostate Cancer Patients Receiving Androgen Deprivation Therapy
Brief Title: The Effect of Multidisciplinary Care Approach on CV Risk Modification in CaP Patients Receiving ADT
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Chi Fai, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2023.509
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Risk; Prostate Cancer
Keywords: Prostate Cancer; Androgen deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCa receiving ADT: prostate cancer patients receiving androgen deprivation therapy

SUMMARY:
Prostate cancer is characterised by its slow progression nature, and even for metastatic disease, the 5-year survival is up to 30%. While ADT can effectively control disease, there is increasing evidence suggesting that it can also result in many adverse cardiovascular side effects on the patients, and these effects are particularly important due to the prolonged survival of these patients. There are suggestions that close cardiovascular (CV) monitoring will help to reduce cardiovascular risk and related morbidities. However, there is limited data to show the positive impact of these monitoring could reducing CV risk and morbidities. Moreover, information regarding the optimal follow-up approach and schedule is also lacking. Therefore, there is a need to have more information on the approach to monitoring the CV risk and the real-life impact of this monitoring on our patients. Patients diagnosed with prostate cancer and plan to receive ADT are invited to participate in this study to assess the potential benefit of multidisciplinary care approach to CV risk modification.

DETAILED DESCRIPTION:
Prostate Cancer (PCa) and androgen deprivation therapy (ADT) PCa is the most common cancer and the second leading cancer death in adult male globally. In Hong Kong, it is one of the most rapidly increasing cancer and is now the third most common cancer and the 4th leading cancer death in male. Despite the increased usage of serum PSA for early cancer diagnosis, more than 50% of patients were diagnosed at stage III & IV, with lymph node +/- bone / visceral metastasis. Therefore, ADT is still commonly used in PCa patients, both as neo-adjuvant/ adjuvant to radiotherapy,as well as backbone therapy for metastatic disease.While the overall survival of PCa patients has been prolonged by ADT, there is also increasing concern about potential long-term side effects, in particular cardiovascular effect.

Therefore, there is a need for prospective studies to understand the role of close cardiovascular assessment, monitoring and treatment on the cardiovascular risk of PCa patients receiving ADT. Information on the risk factors at baseline; follow-up, and also treatment / secondary prevention adopted, will help to provide evidence to fill the current knowledge gap and build practical guidelines for clinical usage. In the long run, the data will also help to estimate the medical resources required for future health care planning to cope with the medical needs of the rapidly increasing PCa population.

ELIGIBILITY:
Inclusion Criteria:

* Adult men 18-80 years old
* With histological proven prostate cancer or clinically diagnosed to have prostate cancer,
* Planned for ADT for at least 1 year

Exclusion Criteria:

* Subjects with established major atherosclerotic cardiovascular disease (ASCVD) as defined by a recent acute coronary syndrome within the past 12 months, a history of myocardial infarction other than the recent acute coronary syndrome event, a history of ischemic stroke, and symptomatic peripheral arterial disease (defined as history of claudication with ankle-brachial index <0.85 or previous revascularization or amputation
* Prior neoadjuvant or adjuvant hormone therapy within 1 year before
* Refuse or unable to give written informed consent
* Participation in an investigational program with interventions outside of routine clinical practice

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patient are eligible as prostate cancer can only develop in males.
Study Population: prostate cancer patients receiving androgen deprivation therapy
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
The change in Framingham Risk Score between baseline and 1-year after ADT. | From enrollment to 1-year after ADT
  The Framingham Risk Score is a gender-specific algorithm based on multiple cardiovascular risk factors including age, smoking status, blood pressure level, serum total cholesterol and HDL-cholesterol level for the estimation of the 10-year risk of developing cardiovascular disease. This remain a commonly used assessment for cardiovascular risk, including PCa patients treated with ADT internationally.

SECONDARY OUTCOMES:
Incidence of new-onset diabetes | From enrollment to 1-year after ADT
  Incidence of new-onset diabetes after ADT
Incidence of new-onset hypertension | From enrollment to 1-year after ADT
  Incidence of new-onset hypertension after ADT
Changes in fasting blood sugar | From enrollment to 1-year after ADT
  Changes in fasting blood sugar (serum level)
Changes in LDL-Cholesterol | From enrollment to 1-year after ADT
  Changes in LDL-Cholesterol (serum level)
Changes in HDL-cholesterol | From enrollment to 1-year after ADT
  Changes in HDL-cholesterol (serum level)
Changes in triglyceride | From enrollment to 1-year after ADT
  Changes in triglyceride (serum level)
Changes in HbA1c | From enrollment to 1-year after ADT
  Changes in HbA1c (serum level)
Incidence of additional medical therapies for optimization of cardiovascular risk | From enrollment to 1-year after ADT
  Number of additional cardiovascular medical therapies
Change in pulse wave velocity | From enrollment to 1-year after ADT
  Change in pulse wave velocity assessed by the Vascular Profiler-1000 machine (Omron, Kyoto, Japan) using the oscillometric cuff technique
Change in Quality of life | From enrollment to 1-year after ADT
  EQ-5D (EuroQol 5 dimensions) questionnaire Quality of life measured by ED-5Q questionnaire, with 5 components [Mobility, Self Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression)], and a Visual analogue scale from 0 to 100 (EQ-VAS) score, the higher the score the better in quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] D'Agostino RB Sr, Vasan RS, Pencina MJ, Wolf PA, Cobain M, Massaro JM, Kannel WB. General cardiovascular risk profile for use in primary care: the Framingham Heart Study. Circulation. 2008 Feb 12;117(6):743-53. doi: 10.1161/CIRCULATIONAHA.107.699579. Epub 2008 Jan 22. PMID 18212285
- [Background] Ghadessi M, Tang R, Zhou J, Liu R, Wang C, Toyoizumi K, Mei C, Zhang L, Deng CQ, Beckman RA. A roadmap to using historical controls in clinical trials - by Drug Information Association Adaptive Design Scientific Working Group (DIA-ADSWG). Orphanet J Rare Dis. 2020 Mar 12;15(1):69. doi: 10.1186/s13023-020-1332-x. PMID 32164754
- [Background] 21. Ng CF, Wei Y, Ong TA, Chan W, Chu PSK, Huang CY, et al. The changes in metabolic profiles and cardiovascular risk in Asian prostate cancer patients after androgen deprivation therapy - a prospective real-life evaluation. Int J Urol 2020; 27 S1: UOP-1430.
- [Background] Ng CF, Teoh JYC, Chiu PKF. Letter by Ng et al Regarding Article, "Cardiovascular Safety of Degarelix Versus Leuprolide in Patients With Prostate Cancer: The Primary Results of the PRONOUNCE Randomized Trial". Circulation. 2022 Mar 22;145(12):e773-e774. doi: 10.1161/CIRCULATIONAHA.121.057407. Epub 2022 Mar 21. No abstract available. PMID 35312383
- [Background] Lopes RD, Higano CS, Slovin SF, Nelson AJ, Bigelow R, Sorensen PS, Melloni C, Goodman SG, Evans CP, Nilsson J, Bhatt DL, Clarke NW, Olesen TK, Doyle-Olsen BT, Kristensen H, Arney L, Roe MT, Alexander JH; PRONOUNCE Study Investigators. Cardiovascular Safety of Degarelix Versus Leuprolide in Patients With Prostate Cancer: The Primary Results of the PRONOUNCE Randomized Trial. Circulation. 2021 Oct 19;144(16):1295-1307. doi: 10.1161/CIRCULATIONAHA.121.056810. Epub 2021 Aug 30. PMID 34459214
- [Background] Narayan V, Ross AE, Parikh RB, Nohria A, Morgans AK. How to Treat Prostate Cancer With Androgen Deprivation and Minimize Cardiovascular Risk: A Therapeutic Tightrope. JACC CardioOncol. 2021 Dec 21;3(5):737-741. doi: 10.1016/j.jaccao.2021.09.014. eCollection 2021 Dec. PMID 34988484
- [Background] Leong DP, Mukherjee SD. The European Society of Cardiology Cardio-Oncology Guidelines: Evidence Base, Actionability, and Relevance to Clinical Practice. JACC CardioOncol. 2022 Dec 6;5(1):137-140. doi: 10.1016/j.jaccao.2022.10.009. eCollection 2023 Feb. No abstract available. PMID 36875915
- [Background] Lyon AR, Lopez-Fernandez T, Couch LS, Asteggiano R, Aznar MC, Bergler-Klein J, Boriani G, Cardinale D, Cordoba R, Cosyns B, Cutter DJ, de Azambuja E, de Boer RA, Dent SF, Farmakis D, Gevaert SA, Gorog DA, Herrmann J, Lenihan D, Moslehi J, Moura B, Salinger SS, Stephens R, Suter TM, Szmit S, Tamargo J, Thavendiranathan P, Tocchetti CG, van der Meer P, van der Pal HJH; ESC Scientific Document Group. 2022 ESC Guidelines on cardio-oncology developed in collaboration with the European Hematology Association (EHA), the European Society for Therapeutic Radiology and Oncology (ESTRO) and the International Cardio-Oncology Society (IC-OS). Eur Heart J. 2022 Nov 1;43(41):4229-4361. doi: 10.1093/eurheartj/ehac244. No abstract available. PMID 36017568
- [Background] Li JKM, Wang LL, Wong CYP, Chiu PKF, Teoh JYC, Kwok HSW, Leung SCH, Wong SH, Tsui SKW, Ng CF. A cross-sectional study on gut microbiota in prostate cancer patients with prostatectomy or androgen deprivation therapy. Prostate Cancer Prostatic Dis. 2021 Dec;24(4):1063-1072. doi: 10.1038/s41391-021-00360-1. Epub 2021 Apr 13. PMID 33850270
- [Background] Teoh JY, Tian XY, Wong CY, Lau CW, Cheng CK, Tang VW, Chan RC, Huang Y, Ng CF. Endothelial dysfunction after androgen deprivation therapy and the possible underlying mechanisms. Prostate. 2022 Jan;82(1):13-25. doi: 10.1002/pros.24244. Epub 2021 Sep 27. PMID 34570375
- [Background] Wong C, Chu P, Teoh J, Chiu P, Yee CH, Chau L, Chan M, Wan H, Leung S, Ng CF. Risks of metabolic diseases and androgen deprivation therapy for prostate cancer in a Chinese population: a prospective multi-centre cohort study. Int Urol Nephrol. 2022 May;54(5):993-1000. doi: 10.1007/s11255-022-03151-2. Epub 2022 Feb 25. PMID 35217907
- [Background] Ng CF, Chiu PKF, Yee CH, Lau BSY, Leung SCH, Teoh JYC. Effect of androgen deprivation therapy on cardiovascular function in Chinese patients with advanced prostate cancer: a prospective cohort study. Sci Rep. 2020 Oct 22;10(1):18060. doi: 10.1038/s41598-020-75139-w. PMID 33093594
- [Background] Chan JSK, Tang P, Hui JMH, Lee YHA, Dee EC, Ng K, Liu K, Tse G, Ng CF. Association between duration of gonadotrophin-releasing hormone agonist use and cardiovascular risks: A population-based competing-risk analysis. Prostate. 2022 Nov;82(15):1477-1480. doi: 10.1002/pros.24423. Epub 2022 Aug 1. PMID 35915869
- [Background] Teoh JY, Chiu PK, Chan SY, Poon DM, Cheung HY, Hou SS, Ng CF. Androgen deprivation therapy, diabetes and poor physical performance status increase fracture risk in Chinese men treated for prostate cancer. Aging Male. 2015;18(3):180-5. doi: 10.3109/13685538.2015.1046043. Epub 2015 May 25. PMID 26004988
- [Background] Teoh JY, Chiu PK, Chan SY, Poon DM, Cheung HY, Hou SS, Ng CF. Risk of new-onset diabetes after androgen deprivation therapy for prostate cancer in the Asian population. J Diabetes. 2015 Sep;7(5):672-80. doi: 10.1111/1753-0407.12226. Epub 2014 Dec 22. PMID 25266491
- [Background] Teoh JY, Chan SY, Chiu PK, Poon DM, Cheung HY, Hou SS, Ng CF. Risk of acute myocardial infarction after androgen-deprivation therapy for prostate cancer in a Chinese population. BJU Int. 2015 Sep;116(3):382-7. doi: 10.1111/bju.12967. Epub 2015 Mar 7. PMID 25327618
- [Background] Teoh JY, Ng CF. Cardiovascular risk after androgen deprivation therapy for prostate cancer: an Asian perspective. Int Urol Nephrol. 2016 Sep;48(9):1429-35. doi: 10.1007/s11255-016-1337-5. Epub 2016 Jun 2. PMID 27256399
- [Background] Levine GN, D'Amico AV, Berger P, Clark PE, Eckel RH, Keating NL, Milani RV, Sagalowsky AI, Smith MR, Zakai N; American Heart Association Council on Clinical Cardiology and Council on Epidemiology and Prevention, the American Cancer Society, and the American Urological Association. Androgen-deprivation therapy in prostate cancer and cardiovascular risk: a science advisory from the American Heart Association, American Cancer Society, and American Urological Association: endorsed by the American Society for Radiation Oncology. Circulation. 2010 Feb 16;121(6):833-40. doi: 10.1161/CIRCULATIONAHA.109.192695. Epub 2010 Feb 1. No abstract available. PMID 20124128
- [Background] Hu JR, Duncan MS, Morgans AK, Brown JD, Meijers WC, Freiberg MS, Salem JE, Beckman JA, Moslehi JJ. Cardiovascular Effects of Androgen Deprivation Therapy in Prostate Cancer: Contemporary Meta-Analyses. Arterioscler Thromb Vasc Biol. 2020 Mar;40(3):e55-e64. doi: 10.1161/ATVBAHA.119.313046. Epub 2020 Jan 23. PMID 31969015
- [Background] Faris JE, Smith MR. Metabolic sequelae associated with androgen deprivation therapy for prostate cancer. Curr Opin Endocrinol Diabetes Obes. 2010 Jun;17(3):240-6. doi: 10.1097/MED.0b013e3283391fd1. PMID 20404727
- [Background] Bolla M, Van Tienhoven G, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Billiet I, Torecilla JL, Pfeffer R, Cutajar CL, Van der Kwast T, Collette L. External irradiation with or without long-term androgen suppression for prostate cancer with high metastatic risk: 10-year results of an EORTC randomised study. Lancet Oncol. 2010 Nov;11(11):1066-73. doi: 10.1016/S1470-2045(10)70223-0. Epub 2010 Oct 7. PMID 20933466
- [Background] Cornford P, Bellmunt J, Bolla M, Briers E, De Santis M, Gross T, Henry AM, Joniau S, Lam TB, Mason MD, van der Poel HG, van der Kwast TH, Rouviere O, Wiegel T, Mottet N. EAU-ESTRO-SIOG Guidelines on Prostate Cancer. Part II: Treatment of Relapsing, Metastatic, and Castration-Resistant Prostate Cancer. Eur Urol. 2017 Apr;71(4):630-642. doi: 10.1016/j.eururo.2016.08.002. Epub 2016 Aug 31. PMID 27591931
- [Background] 1. Hong Kong Cancer registry - Prostate cancer in 2020 https://www3.ha.org.hk/cancereg/pdf/factsheet/2020/prostate_2020.pdf
- [Background] Leong DP, Fradet V, Shayegan B, Duceppe E, Siemens R, Niazi T, Klotz L, Brown I, Chin J, Lavallee L, Mousavi N, Luke P, Lukka H, Gopaul D, Violette P, Hamilton RJ, Davis MK, Karampatos S, Mian R, Delouya G, Fradet Y, Mukherjee S, Conen D, Chen-Tournoux A, Johnson C, Bessissow A, Dresser G, Hameed AK, Abdel-Qadir H, Sener A, Pal R, Devereaux PJ, Pinthus J. Cardiovascular Risk in Men with Prostate Cancer: Insights from the RADICAL PC Study. J Urol. 2020 Jun;203(6):1109-1116. doi: 10.1097/JU.0000000000000714. Epub 2020 Jan 3. PMID 31899651